CLINICAL TRIAL: NCT01049620
Title: A Phase I Dose Finding Study of RAD001 in Combination With Capecitabine and Oxaliplatin (XELOX) in Patients With Advanced Gastric Cancer
Brief Title: RAD001 in Combination With Capecitabine and Oxaliplatin (XELOX) in Patients With Advanced Gastric Cancer: RAD001+XELOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0905
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
Keywords: XELOX; RAD001; phase 1
MeSH Terms: interventions — Everolimus; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xelox+RAD001 (Experimental)
  Interventions: Drug: RAD001, Capecitabine, Oxaliplatin

INTERVENTIONS:
Drug: RAD001, Capecitabine, Oxaliplatin — Dose level -1 : Capecitabine 800mg/m2 po bid D1-14, Oxaliplatin 100mg/m2 iv D1 RAD001 5mg po qd D1-21
  Dose level 1 : Capecitabine 800mg/m2 po bid D1-14, Oxaliplatin 100mg/m2 iv D1 RAD001 7.5mg po qd D1-21
  Dose level 2 : Capecitabine 800mg/m2 po bid D1-14, Oxaliplatin 130mg/m2 iv D1 RAD001 7.5mg po qd D1-21
  Dose level 3 : Capecitabine 1000mg/m2 po bid D1-14, Oxaliplatin 100mg/m2 iv D1 RAD001 7.5mg po qd D1-21
  Dose level 3A : Capecitabine 800mg/m2 po bid D1-14, Oxaliplatin 130mg/m2 iv D1 RAD001 10mg po qd D1-21
  Dose level 3B : Capecitabine 1000mg/m2 po bid D1-14, Oxaliplatin 100mg/m2 iv D1 RAD001 10mg po qd D1-21
  Dose level 4 : Capecitabine 1000mg/m2 po bid D1-14, Oxaliplatin 130mg/m2 iv D1 RAD001 7.5mg po qd D1-21
  Dose level 5 : Capecitabine 1000mg/m2 po bid D1-14, Oxaliplatin 130mg/m2 iv D1 RAD001 10mg po qd D1-21

SUMMARY:
It is expected that RAD001 works in gastric cancer by inhibiting PI3K/AKT/mTOR pathway and Hif1A (hypoxia inducible factor 1, alpha subunit), a key player in angiogenesis and the growth of tumors like renal cell carcinoma.However, RAD001 alone looks not enough to control gastric cancer. By the mechanisms above, RAD001 can show additive or synergistic effect in combination with conventional chemotherapy. In this study, XELOX was selected as a conventional combination chemotherapy because it was proven very active and safe in gastric cancer. Combination of XELOX and RAD001 has been never tried for the treatment of cancer patients yet. So, the optimal dose will be first determined in this phase I study

DETAILED DESCRIPTION:
For the first cohort of this phase I study, each drug of capecitabine, oxaliplatin, and RAD001 will be started at one or two dose below the ordinary full dose of each drug as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented unresectable or metastatic adenocarcinoma of stomach or gastroesophageal junction
* No history of chemotherapy or radiation
* Age 18 to 70 years old
* Estimated life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow function (white blood cell counts >3,000/uL, absolute neutrophil count>1,500/uL, Platelets>100,000/uL, Hgb>8 g/dL)
* Adequate kidney function (creatinine<1.5 mg/dL)
* Adequate liver function (bilirubin<1.5 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level <3 times the upper normal limit (5 times for patients with liver metastasis))
* Signed written informed consent

Exclusion Criteria:

* Past or concurrent history of neoplasm other than gastric adenocarcinoma except for curatively treated basal cell carcinoma of skin or in situ carcinoma of the cervix uteri
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start
* Presence of central nervous system metastasis
* Bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Peripheral neuropathy (NCI CTC AE version 3.0 > Grade I)
* History of significant neurologic or psychiatric disorders
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions
* Patients with known history of ischemic heart disease and/or with myocardial infarction
* Known allergy to study drugs
* Administration of drugs showing interaction with RAD001

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose (MTD) | 1year

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Overall survival | 1 year
Biomarker study | 1 year
Response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea